CLINICAL TRIAL: NCT01518959
Title: Phase III, Controlled, Double-blind, Randomized Study of 25-OH-Vitamin-D3 Substitution in Patients With Malignant and Immune-hematologic Diseases
Brief Title: The Effect of 25-OH-Vitamin-D3 Substitution in Patients With Malignant and Immune-hematologic Diseases
Acronym: D-HEM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment rate; technical issues with sample storage
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Istvan Takacs, Clinical Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-HEM
Record Dates: First submitted 2012-01-06; First posted 2012-01-26 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Chronic Lymphoid Leukemia
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): no treatment
  Interventions: Drug: oleum neutralicum
- Cholecalcipherol (Active Comparator): Treatment with 180 000 IU cholecalcipherol monthly
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 180.000 IU monthly
  Arms: Cholecalcipherol
Drug: oleum neutralicum — Placebo comparator, 9 ml monthly
  Arms: Placebo

SUMMARY:
Recent data have shown that the inadequate vitamin D status plays a role in the manifestation of the haematologic tumors and serum vitamin D level has a prognostic role also as it determines the tumor mortality. But data have not proved a causal relationship between the inadequate vitamin D status and the unfavourable outcomes so far. It is also still unknown, whether the normalization of vitamin D status in patient with vitamin D inadequacy is able to improve the prognosis and survival.

In this study the investigators examine the role of the adequate vitamin D substitution in the improvement of the outcomes of haematologic disorders.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old male or female
* chronic lymphoid leukaemia, any Rai stage
* 25-OH-Vitamin-D3 level between 10 and 30 ng/mL

Exclusion Criteria:

* serum calcium > 2,60 mmol/l
* 24 hour calcium urine excretion > 0,1 mmol/kg/day
* serum phosphate > 1,45 mmol/l
* eGFR < 30 ml/min/1,73m2
* nephrolithiasis
* receiving parenteral vitamin-D3 in past 6 months
* activated vitamin-D3 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 5 years

SECONDARY OUTCOMES:
Time to treatment needed | up to 5 years
Blood lymphocyte count | monthly, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Takacs, MD, PhD, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University - 1st Departement of Internal Medicine, Budapest, Hungary